CLINICAL TRIAL: NCT05553080
Title: Significance of Immunohistochemical Expression of Fascin-1 in Colorectal Carcinoma
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, Lecturer of Pathology, Sohag University
Other Study IDs: Soh-Med-22-09-14
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-10

CONDITIONS: Cancer of Colon
Keywords: Cancer Colon; Fascin-1; Actin assembly
MeSH Terms: conditions — Colonic Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Immunohistochemistry — immunohistochemical staining of colorectal carcinoma specimens by anti human fascin antibody.

SUMMARY:
Colorectal carcinoma is a major health problem. As a malignant tumor, the malignant potential of colorectal carcinoma is based mainly on its ability to metastasis to different sites. Fascin-1 is an actin binding protein which is involved in reconstruction of intracellular actin network, the latter enforces the neoplastic cell to invade surrounding structures.

DETAILED DESCRIPTION:
colorectal carcinoma is an aggressive malignant tumor. It has high incidence of cancer-related morbidity and mortality. the malignant potential of a given neoplasm is based mainly on its ability to invade the surrounding vasculature and reach to distant sites, the latter is called metastasis. in order to metastasize to distant sites, the neoplastic cells must re-arrange the intracellular actin filaments into well formed intracellular assembly which enable the neoplastic cells to reach to distant sites. Fascin-1 is an actin binding protein, it is involved in reconstruction of actin assembly. fortunately, Fascin-1 could be blocked by newly developed medications, blocking of Fascin-1 may limit the metastasis of colorectal carcinoma. in current study the investigators detect Fascin-1 in colorectal carcinoma by immunohistochemical approach, then they correlated different levels of Fascin-1 expression to tumor clinical and pathological criteria as patients' ages, sexes, tumor stages, nodal metastasis, vascular and per-ineural invasions.

ELIGIBILITY:
Inclusion Criteria:

* All cases of colorectal carcinoma.

Exclusion Criteria:

* cases diagnosed on basis of lower endoscopic biopsies or local resections without radical colectomy.
* Patients with preopoerative history of chemo or radiotherapy.
* Patients with poor clinical data.

Ages: 30 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients had colorectal carcinoma who underwent radical colectomy operations in Sohag University Hospital, Sohag, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of immunohistochemical staining of colorectal carcinoma by Fascin-1 | September , 2022
  correlation of different levels of Fascin-1 expression to patients' ages, sexes, tumor stage, nodal metastasis, vascular and perineural invasion.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Maisa Hashem Mohammed, Sohag
  - Sohag faculty of medicine, Sohag

IPD SHARING:
Plan to Share IPD: Undecided